CLINICAL TRIAL: NCT02969135
Title: Physiotherapy With Progressive Active Exercise Training After Surgical Rotator Cuff Repair -A Randomized Controlled Trial With 3 and 12 Months Follow-up
Brief Title: Progressive Active Exercise After Surgical Rotator Cuff Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marius Henriksen (Other)
Responsible Party: Sponsor-Investigator, Marius Henriksen, Professor, Frederiksberg University Hospital
Organization: Frederiksberg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FYS012
Record Dates: First submitted 2016-11-15; First posted 2016-11-21 (Estimated); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Rotator Cuff Tear
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive early passive and active movement (Experimental): Active exercise starts one week after surgery.
  Interventions: Behavioral: Progressive early passive and active movement
- Limited early passive movement (Active Comparator): Active exercise starts six weeks after surgery.
  Interventions: Behavioral: Limited early passive movement

INTERVENTIONS:
Behavioral: Progressive early passive and active movement — Post-surgical physical therapy including active exercise
  Arms: Progressive early passive and active movement
Behavioral: Limited early passive movement — Post-surgical physical therapy including passive mobilisation
  Arms: Limited early passive movement

SUMMARY:
Shoulder disorders are extremely common, with a life-time prevalence in population of 30%. About 23% of the working population with shoulder problems are sick-listed. Specifically rotator cuff tears are considered some of the principal causes of chronic shoulder pain and disability, especially with advancing age. The National Patient Register in Denmark has registered 730 rotator cuff repairs in 2006 and 990 in 2012, which represents a 35% increase.

A rotator cuff tear is defined as a rupture of the tendon (s) of the shoulder, and most frequently involves the supraspinatus and/or the infraspinatus tendon, resulting in loss of function due to pain and tissue weakness. Little is known about the effects of the postoperative training/rehabilitation, and this provides an unclear picture of the total treatment procedure of this condition.

The Danish National Clinical Guidelines from 2013 recommend that these patients are offered rehabilitation and that the shoulder is immobilized post-surgery, but the evidence for postoperative training is moderate- low. The past few years, there have been conducted 5 systematic reviews looking at different rehabilitation parameters after rotator cuff surgery. They conclude that early Range-Of-Motion exercise accelerate healing, reduce stiffness, do not increase risk of re-rupture and that immobilization do not increase tendon healing or clinical outcome. They also conclude that there is a further need to evaluate approaches that foster early initiation of rehabilitation and gradual introduction of functional load in high-quality, adequately powered trials, also considering key outcomes such as return to work.

Therefore, the aim of this study is to compare the effect of a progressive early passive and active movement protocol with a care as usual (limited early passive movement protocol) on tendon healing, physical function, pain, and quality of life, in patients operated due to traumatic full thickness rotator cuff tear in a Randomized Controlled Trial.

Shortterm effects of physical function, pain, and quality of life will be studied as primary patient reported outcome, while secondary outcomes will be clinical and paraclinical outcomes in addition to the longterm effects of physical function, pain, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Women and men above 18 years
* Operated due to traumatic full thickness RC-tear
* Involving supraspinatus (full thickness and width)
* Present with reduced arm elevation strength and pain
* Clinical diagnosis verified by arthroscopy
* Fully repairable RC-tear

Exclusion Criteria:

* Patients with non-traumatic RC-tears of the shoulder
* Patients with isolated teres minor or subscapularis tear
* Patients with partial thickness/ width tear
* Prior shoulder surgery (all shoulder joints)
* Glenohumeral osteo arthrosis (OA), rheumatoid arthritis or periarthrosis
* Inability to speak or read Danish
* Inability to perform and maintain the physical training
* Other condition negatively influencing compliance or conditions that in the opinion of the investigator puts a potential participant at increased risk or otherwise makes him/her unsuitable for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2017-02-26 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-05-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Western Ontario Rotator Cuff Index (WORC) | 12 weeks

SECONDARY OUTCOMES:
Change from baseline in Western Ontario Rotator Cuff Index (WORC) | 6 and 52 weeks
Change from baseline in Disability Arm Shoulder Hand (DASH) | 6, 12 and 52 weeks
Global Rating Scale (GRS) | 6, 12 and 52 weeks
  Global perceived treatment effect
Change from baseline in Numeric Pain Rating Scale (NPRS) | 6, 12 and 52 weeks
Change from baseline in Shoulder Range of Motion (ROM) | 6, 12 and 52 weeks
Change from baseline in Shoulder Muscle Strength (maximum isometric voluntary contraction) of external and internal rotation and scaption | 12 and 52 weeks
  Maximum isometric voluntary contraction (MVC) of external and internal rotation and scaption (elevation in scapular plane) measured by IsoForce EVO2 dynamometer.

OTHER OUTCOMES:
Ultrasound imaging of rotator cuff tendons | 6 weeks
  Assessment of possible re-ruptures of tendons
Ultrasound Imaging of rotator cuff tendons | 52 weeks
  Tendon healing characteristics of the repaired tendon compared to the healthy shoulder tendons
Return to work | 6 and 52 weeks
  Patient-reported time (days) til return to full work capacity.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Bispebjerg and Frederiksberg Hospitals, Copenhagen
  - Herlev and Gentofte Hospital, Copenhagen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kjaer BH, Svensson RB, Warming S, Peter Magnusson S. Supraspinatus Muscle and Tendon Characteristics 1 Year After Surgical Rotator Cuff Repair Compared With Contralateral Shoulder: Data From the CUT-N-MOVE Trial. Am J Sports Med. 2024 Jul;52(8):2082-2091. doi: 10.1177/03635465241255143. Epub 2024 Jun 11. PMID 38860727
- [Derived] Kjaer BH, Magnusson SP, Henriksen M, Warming S, Boyle E, Krogsgaard MR, Al-Hamdani A, Juul-Kristensen B. Effects of 12 Weeks of Progressive Early Active Exercise Therapy After Surgical Rotator Cuff Repair: 12 Weeks and 1-Year Results From the CUT-N-MOVE Randomized Controlled Trial. Am J Sports Med. 2021 Feb;49(2):321-331. doi: 10.1177/0363546520983823. Epub 2021 Jan 20. PMID 33471547
- [Derived] Kjaer BH, Magnusson SP, Warming S, Henriksen M, Krogsgaard MR, Juul-Kristensen B. Progressive early passive and active exercise therapy after surgical rotator cuff repair - study protocol for a randomized controlled trial (the CUT-N-MOVE trial). Trials. 2018 Sep 3;19(1):470. doi: 10.1186/s13063-018-2839-5. PMID 30176943